CLINICAL TRIAL: NCT04961684
Title: Clinical Evaluation of Efficacy and Safety of a Medical Device for the Treatment of Toenail Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19E2407
Record Dates: First submitted 2021-05-31; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Onychomycosis of Toenail

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solver Pen (Experimental)
  Interventions: Device: Solver Pen
- Loceryl 5% (Active Comparator)
  Interventions: Drug: Loceryl 5%

INTERVENTIONS:
Device: Solver Pen — One application per day for 3 months
  Arms: Solver Pen
Drug: Loceryl 5% — One application per week for 3 months
  Arms: Loceryl 5%

SUMMARY:
The efficacy and safety of Solver Pen (prototype number X92001704) is evaluated in this randomized, open label, controlled, investigator-blinded, comparative clinical trial in 76 patients. Subjects are treated with either the test medical device (Solver Pen) or the comparator (Loceryl, 5% amorolfine), respectively, for a period of 90 days. The primary objective of the investigation is the increase of percentage of healthy surface on the great toenail at study end versus baseline, as evaluated by a blinded investigator. Patients are followed up for a period of 90 days, with visits at D0 (baseline), D30, D60 and D90, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patient having given her/his informed, written consent.
2. Patient cooperative and aware of the modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.
3. Patient being psychologically able to understand information and to give their/his/her consent.
4. Age: more than 18 years.
5. Subject with superficial onychomycosis on at least one great toenail or light to moderate disto-lateral onychomycosis (without matrix involvement and involvement <2/3 of the tablet).
6. Patient with positive KOH staining.
7. Patient having stopped any systemic antifungal treatment since at least 6 months before inclusion and/or any topical antifungal treatment since at least 3 months before inclusion.
8. Women of childbearing potential should use an accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after study end.

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the investigation;
2. Patient considered by the Investigator likely to be non-compliant with the protocol.
3. Patient enrolled in another clinical trial during the test period.
4. Subject having a known allergy to one of the constituents of the tested products.
5. Patient with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk;
6. Patient suffering from serious or progressive diseases (to investigator's discretion) such as uncontrolled diabetes, peripheral circulatory disease, HIV, psoriasis, lichen planus, immunosuppressive pathology…
7. Subject with cutaneous pathology on studied zone (other than onychomycosis like angioma, dermatitis…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Percentage of healthy surface (performance) | 90 days
  Variation of the percentage of healthy surface after 90 days of treatment with the test medical device or reference versus baseline value. Evaluation is done in blind by digital analysis of photographs of the great, infected toenail.

SECONDARY OUTCOMES:
Percentage of healthy surface (performance) | 30 and 60 days
  Variation of the percentage of healthy surface after 30 and 60 days of treatment with the test medical device or reference versus baseline. Blinded evaluation is performed by digital analysis of photographs of the great, infected toenail.
Microbiological efficacy: KOH staining (performance) | 90 days
  Evaluation of microbiological efficacy of both treatments by KOH staining on D90 versus baseline.
Microbiological efficacy: fungal culture (performance) | 90 days
  Evaluation of microbiological efficacy of both treatments by fungal culture on D90 versus baseline.
Clinical efficacy: onychomycosis evolution (performance) | 30, 60 and 90 days
  Blinded assessment of clinical efficacy of both treatments on D0 (baseline), D30, D60 and D90 by evaluation of onychomycosis evolution on a 4-point scale (failure to success)
Clinical efficacy: onycholysis (performance) | 30, 60 and 90 days
  Blinded assessment of clinical efficacy of both treatments on D0 (baseline), D30, D60 and D90 by evaluation of onycholysis on a 5-point scale (none to severe)
Clinical efficacy: nail distrophy (performance) | 30, 60 and 90 days
  Blinded assessment of clinical efficacy of both treatments on D0 (baseline), D30, D60 and D90 by evaluation of nail distrophy on a 5-point scale (none to severe)
Clinical efficacy: nail discoloration (performance) | 30, 60 and 90 days
  Blinded assessment of clinical efficacy of both treatments on D0 (baseline), D30, D60 and D90 by evaluation of nail discoloration on a 5-point scale (none to severe)
Clinical efficacy: nail thickening (performance) | 30, 60 and 90 days
  Blinded assessment of clinical efficacy of both treatments on D0 (baseline), D30, D60 and D90 by evaluation of nail thickening on a 5-point scale (none to severe)
Impact on quality of life (performance) | 60 and 90 days
  Evaluation of the impact on the quality of life (QoL) of the patients using a validated questionnaire (NailQoL: Nail Questionnaire Of Life from 0=no impact on life quality to 100=maximum impact on life quality) before (baseline) and 60 and 90 days of treatment with the test medical device or reference, respectively.
Subjective evaluation questionnaire for the patient (performance) | 14, 30, 60 and 90 days of treatment
  Evaluation of efficacy, tolerance, and acceptability cosmetic aspect, usability…) of the investigational device by the patients using a subjective evaluation questionnaire (answers to questions with 5 modalities from "strongly disagree" to "strongly agree"), performed at each visit and at D14 (via phone).
Assessment of local tolerance by the investigator (safety and tolerability) | 30, 60 and 90 days
  Evaluation of local tolerance of the test medical device at each visit. Assessment is performed by the investigator via clinical evaluation and subject interrogation on a scale from 0 (bad tolerance) to 3 (very good tolerance)
Incidence of Adverse events (safety and tolerability) | 30, 60 and 90 days
  Collection of Adverse events and adverse device effects throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Nejib Doss, MD, Principal Investigator — Eurofins Dermscan Tunisia
Locations (1):
- Pr Doss office, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No